CLINICAL TRIAL: NCT02919423
Title: TMS Modulation of Insula-related Brain Networks.02
Acronym: TMSINS02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00077293
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 Hz TMS (Active Comparator): active TMS will be administered
  Interventions: Device: transcranial magnetic stimulation
- 1 Hz TMS (Active Comparator): active TMS will be administered
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation

SUMMARY:
The purpose of this study is to investigate the modulatory effects of repetitive transcranial magnetic stimulation (rTMS) on functional connectivity with the insula. Functional connectivity (FC) measures the interaction between brain regions, and recent neuroimaging studies have used FC to investigate how addiction affects FC among pertinent brain regions. rTMS, which can excite cortical neurons, has shown promise as a method to manipulate brain connectivity and could be used therapeutically to treat addiction. However, investigators first need more information on brain FC and how it relates to behavior, in order to guide rTMS target selection.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* between the ages of 18-55
* right-handed

Exclusion Criteria:

* significant health problems (e.g., current and uncontrolled liver, lung, or heart problems) or presence of medical illness likely to alter brain morphology (including history of seizure, history of epilepsy in self or first degree relatives, stroke, brain surgery, head injury, and known structural brain lesion)
* current diagnosis of Axis I psychiatric disorders (e.g., depression, anxiety disorder, schizophrenia)
* meet DSM-5 criteria for current substance use disorder other than nicotine
* use of psychoactive medications that would result in a positive urine drug screen
* Current use of medications known to lower the seizure threshold
* positive breath alcohol concentration
* presence of conditions that would make MRI unsafe (e.g., metal implants, pacemakers)
* among women, a positive urine pregnancy test
* vision that cannot be corrected to 20/40

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12; Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merideth Addicott, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 subjects were consented but did not meet eligibility criteria and were not randomized to a condition.
Groups:
- 10 Hz TMS: This group received 10 Hz TMS
- 1 Hz TMS: This group received 1 Hz TMS
Period: Overall Study
Arm/Group | 10 Hz TMS | 1 Hz TMS
Started | 6 | 25
Completed | 4 | 16
Not Completed | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 Hz TMS | 1 Hz TMS | Total
Number analyzed (Participants) | 6 | 25 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (7) | 31 (12) | 30 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 18 | 21
  Male | 3 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 7 | 7
  White | 5 | 14 | 19
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 25 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Connectivity Strength Measured With Functional Magnetic Resonance Imaging
Description: Difference in functional connectivity from the TMS target site to the right insula. The primary dependent variable was the resting-state functional connectivity strength between the TMS target site and the right insula.
Time Frame: baseline and 1 week
Measure: Number; unit: correlation coefficient
Arm/Group | 10 Hz TMS | 1 Hz TMS
Number analyzed (Participants) | 6 | 25
correlation coefficient | .25 | .13

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 10 Hz TMS | 1 Hz TMS
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/25
Other Adverse Events (participants affected / at risk) | 0/6 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT02919423/Prot_SAP_000.pdf